CLINICAL TRIAL: NCT02437604
Title: An Open-Label, Crossover Study to Determine the Pharmacokinetic Profile and Tolerability of Single Doses of High Strength Fluticasone Propionate Multidose Dry Powder Inhaler and Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler Compared to High Strength FLOVENT® DISKUS® and ADVAIR® DISKUS® in Patients With Persistent Asthma 12 Years of Age and Older
Brief Title: Study to Determine the Pharmacokinetics and Tolerability of Fluticasone Propionate MDPI and Fluticasone Propionate/Salmeterol MDPI Compared to High Strength FLOVENT® DISKUS® and ADVAIR® DISKUS® in Patients With Persistent Asthma 12 Years of Age and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSS-AS-10042
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Fp MDPI 200 mcg, 1 inhalation
  Interventions: Drug: Treatment A: Fp MDPI
- Treatment B (Experimental): FS MDPI 200/12.5 mcg, 1 inhalation
  Interventions: Drug: Treatment B: FS MDPI
- Treatment C (Active Comparator): fluticasone propionate (FLOVENT DISKUS) 250 mcg, 2 inhalations
  Interventions: Drug: Treatment C Flovent
- Treatment D (Active Comparator): fluticasone propionate/salmeterol (ADVAIR DISKUS) 500/50 mcg, 1 inhalation
  Interventions: Drug: Treatment D: Advair

INTERVENTIONS:
Drug: Treatment A: Fp MDPI — Fp MDPI 200 mcg, 1 inhalation
  Other Names: fluticasone propionate
  Arms: Treatment A
Drug: Treatment B: FS MDPI — FS MDPI 200/12.5 mcg, 1 inhalation
  Other Names: fluticasone propionate/salmeterol
  Arms: Treatment B
Drug: Treatment C Flovent — FLOVENT DISKUS 250 mcg, 2 inhalations
  Other Names: fluticasone propionate
  Arms: Treatment C
Drug: Treatment D: Advair — ADVAIR DISKUS 500/50 mcg, 1 inhalation
  Other Names: fluticasone propionate/salmeterol
  Arms: Treatment D

SUMMARY:
Each patient will participate in the study for approximately 7 weeks. Participation will include a screening period of up to 21 days and 4 treatment periods; each consisting of a 3-day/2-night inpatient period.

ELIGIBILITY:
* Criteria: • Inclusion Criteria:
* The patient has persistent asthma.
* To meet current asthma therapy requirements patients must be currently treated with inhaled corticosteroids (ICSs) at a dose that has been stable for at least 30 days before the SV.
* Written informed consent/assent is obtained. For adult patients (aged 18 years and older, or as applicable per local regulations), the written ICF must be signed and dated by the patient before conducting any study-related procedure. For minor patients (aged 12 to 17 years, or as applicable per local regulations), the written ICF must be signed and dated by the parent/legal guardian and the written assent form must be signed and dated by the patient (if applicable) before conducting any study related procedure. Note: Age requirements are as specified by local regulations.
* The patient is a male or female 12 years of age or older, as of the visit when the ICF/assent form is signed (SV).
* Asthma diagnosis: The patient has a diagnosis of asthma as defined by the NIH. The asthma diagnosis has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in asthma medication) for at least 30 days before providing informed consent.
* The patient is able to demonstrate acceptable and reproducible inhalation technique with the DISKUS device and the Teva MDPI device.
* The patient is able to withhold (as judged by the investigator) his or her rescue medication for at least 6 hours before the SV and before all treatment visits where spirometry is performed.
* The patient has a body mass index (BMI = weight [kg] ÷ height2 [m]) within the 5th and 97thpercentiles for the patient's age and gender. The patient must have a weight of 115 pounds or higher.
* The patient/parent/legal guardian/caregiver is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (eg, dose schedules, visit schedules, blood draws, procedures, and record keeping).

  * Other criteria may apply, please contact the investigator for more information.
* Exclusion Criteria:
* The patient has a history of a life-threatening asthma exacerbation that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the patient's last study-related visit (for eligible patients only, if applicable). Eligible female patients unwilling to employ appropriate contraceptive measures to ensure that pregnancy will not occur during the study will be excluded. Any patient becoming pregnant during the study will be withdrawn from the study.
* The patient has participated as a randomized patient in any investigational drug study within 30 days (starting from the final follow-up visit of that study) preceding the SV or plans to participate in another investigational drug study at any time during this study.
* The patient has previously participated in an Fp MDPI or FS MDPI study. Participation is defined as randomization to treatment.
* The patient has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the study drug (ie, lactose).
* The patient has been treated with any known cytochrome P450 (CYP) 3A4 inhibitors (eg, azole antifungals, ritonavir, or clarithromycin) within 30 days before the SV or plans to be treated with any CYP3A4 inhibitor during the study.The patient has been treated with any of the prohibited medications during the prescribed (per protocol) washout periods before the SV.
* The patient has either lost or donated ≥500 mL of whole blood within the 60 days before the first dose of study drug or the patient has received or donated plasma, white blood cells, or platelets within the 14 days before the first dose of study drug. Patients that have plans to donate blood or blood products during the study or within the 90 days after completion of the study are also excluded.
* The patient currently smokes or has a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient may not have used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco).
* The patient has a culture-documented or suspected bacterial or viral upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI),
* The patient has a history of alcohol or drug abuse within 2 years preceding the SV.
* The patient has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV, or has had any hospitalization for asthma within 2 months before the SV.
* The patient has untreated oral candidiasis at the SV. Patients with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the study. Note: Azole antifungals are prohibited.
* The patient is either an employee or an immediate relative of an employee of the investigational center.
* A member of the patient's household is participating in the study at the same time. However, after the enrolled patient completes or discontinues participation in the study, another patient from the same household may be screened.
* The patient has a disease/condition that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

  * Other criteria may apply, please contact the investigator for more information.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
AUC0-t Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours After administration
Cmax Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours After administration

SECONDARY OUTCOMES:
AUC0-∞ Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
AUC%extrap Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
tmax Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
t½ Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
λz Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
CL/F Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration
Vz/F Plasma drug concentration | 0.08, 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 24, 30, and 36 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (3):
- United States (3):
  - Teva Investigational Site 13178, Raleigh, North Carolina
  - Teva Investigational Site 13177, Edmond, Oklahoma
  - Teva Investigational Site 13179, San Antonio, Texas

REFERENCES:
- [Derived] Nugent C, Yiu G, Song S, Caracta C. The pharmacokinetics, safety, and tolerability of single, high-strength doses of fluticasone propionate and fluticasone propionate/salmeterol delivered via a novel multidose dry powder inhaler in adolescents and adults with persistent asthma. J Asthma. 2018 Aug;55(8):898-906. doi: 10.1080/02770903.2017.1373392. Epub 2017 Oct 30. PMID 28933971